CLINICAL TRIAL: NCT04063098
Title: Effects of Endoscopic Sleeve Gastroplasty on Hormonal Markers of Glucose-homeostasis
Brief Title: Glucose-homeostasis After Endoscopic Sleeve Gastroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ESG_01
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Other): Participants scheduled for endoscopic sleeve gastroplasty
  Interventions: Other: Oral glucose tolerance test

INTERVENTIONS:
Other: Oral glucose tolerance test — Oral glucose tolerance test (OGTT) after a 72-hours standardized diet. OGTT will be performed 1 month prior to as well as 1, 3, 6, and 12 months after endoscopic sleeve gastroplasty

SUMMARY:
Endoscopic sleeve gastroplasty (ESG) is a transoral endoscopic procedure that creates a tubular sleeve along the lesser curvature with a gastric volume of approximately 30%. Summarizing the available literature published since its introduction in 2013, ESG was capable to achieve > 10% of sustained total body weight loss in a majority of mildly to moderately obese patients with the caveat of only minor adverse events. Besides weight loss, little is known about the metabolic effects of ESG. The present study seeks to measure markers of glucose homeostasis during oral glucose tolerance tests before and subsequently after application of ESG in 12 patients.

DETAILED DESCRIPTION:
Endoscopic sleeve gastroplasty (ESG) is a transoral endoscopic procedure that utilizes full-thickness sutures extending from the prepyloric antrum to the gastroesophageal junction, creating a tubular sleeve along the lesser curvature with a gastric volume of approximately 30%. After the first feasibility study was available in 2013, multiple investigators published data on safety and efficacy of ESG. A recent meta analysis of novel endoscopic procedures revealed four observational studies on ESG. At 6, 12 and 24 months pooled excessive weight loss (EWL) was 52%, 53%, and 60% while pooled total body weight loss (TBWL) was 16%, 17%, and 20%, respectively.

Aside from its efficacy in terms of body weight loss, only a small number of investigations addressed metabolic changes in response to ESG so far. In a large retrospective analysis, which observed the outcomes of 1000 patients following ESG, 13 of 17 cases of type 2 diabetes mellitus (T2DM), all 28 cases of hypertension, and 18 of 32 cases of dyslipidemia were in complete remission by the third month of follow-up.

Summarizing the available literature, knowledge about effects of ESG on metabolism and glucose homeostasis is scarce. Available studies are subject to significant limitations in terms of sample size and or generalizability of results. The present study aims at a comprehensive determination of changes in hormonal regulators of glucose homeostasis after ESG in comparison to the preoperative state. Up to date, there are no structured and detailed analyses available that investigate glucose homeostasis following ESG. Proper glucose homeostasis yields a significant impact on a patients' quality of life and may - if deteriorated - be accompanied by a plethora of somatic and psychological constraints. The results of the present study seeks to investigate glucose homeostasis following ESG in detail. This may help to identify patients in need for further assistance regarding their post-interventional lifestyle in order to avoid e.g. hypoglycemia, and to further characterize patients' cohorts that will likely benefit from ESG.

ELIGIBILITY:
Inclusion Criteria:

* Planned ESG
* Written informed consent
* Male or female sex
* Age 18-65 years
* BMI ≥ 40 kg/m2 OR
* BMI ≥ 35 kg/m2 and obesity-related comorbidities except type 2 diabetes

Exclusion Criteria:

* Type 1 or Type 2 Diabetes
* Type 2 Diabetes according to pathological OGTT at visit 2
* Mandatory use of medical drugs that influence glucose metabolism
* Participant had bariatric procedures other than ESG
* Abdominal surgery influencing glucose metabolism
* Moderate to severe chronic kidney, liver, or pancreatic disease
* Pregnancy or breastfeeding
* Physical or psychological disease likely to interfere with the normal conduct of the study and interpretation of the study results as judged by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-05-09 (Actual)

PRIMARY OUTCOMES:
Area under the curve for plasma glucose in oral glucose tolerance test | From time-point 0 to 120 minutes during oral glucose tolerance test, measurement every 15 minutes
  Plasma glucose will be measured in oral glucose tolerance test following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.

SECONDARY OUTCOMES:
Area under the curve for glucagon-like peptide I in oral glucose tolerance test | From time-point 0 to 120 minutes during oral glucose tolerance test, measurement every 15 minutes
  Glucagon-like peptide I will be measured in oral glucose tolerance test following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.
Area under the curve for gastric inhibitory peptide in oral glucose tolerance test | From time-point 0 to 120 minutes during oral glucose tolerance test, measurement every 15 minutes
  Gastric inhibitory peptide will be measured in oral glucose tolerance test following dapagliflozin and will be compared with concentrations measured following placebo. Active and inactivated glucagon like peptide I will be measured.
Area under the curve for glucagon in oral glucose tolerance test | From time-point 0 to 120 minutes during oral glucose tolerance test, measurement every 15 minutes
  Glucagon will be measured in oral glucose tolerance test
Area under the curve for somatostatin in oral glucose tolerance test | From time-point 0 to 120 minutes during oral glucose tolerance test, measurement every 15 minutes
  Somatostatin will be measured in oral glucose tolerance test
Area under the curve for non-acyl ghrelin in oral glucose tolerance test | From time-point 0 to 120 minutes during oral glucose tolerance test, measurement every 15 minutes
  Non-acyl Ghrelin will be measured in oral glucose tolerance test
Area under the curve for insulin in oral glucose tolerance test | From time-point 0 to 120 minutes during oral glucose tolerance test, measurement every 15 minutes
  Insulin will be measured in oral glucose tolerance test

CONTACTS AND LOCATIONS:
Overall Officials: Markus Laimer, Prof. MD, Principal Investigator — Department of Diabetes, Endocrinology, Clinical Nutrition and Metabolism, University Clinics Bern, Inselspital, Bern, Switzerland
Locations (1):
- Department of Diabetes, Endocrinology, Nutritional Medicine and Metabolism, Inselspital, Bern University Hospital, University of Bern, Bern, Switzerland, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: July 30th 2022
Access Criteria: Contact with the Study Sponsor